CLINICAL TRIAL: NCT01651988
Title: EFFICACY OF KETAMINE-PROPOFOL COMBINATION FOR SHORT SURGICAL PROCEDURES
Brief Title: Efficacy of Ketamine-Propofol for Short Surgical Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Cartagena (Other)
Responsible Party: Principal Investigator, Dr. Ricardo Poveda Jaramillo, Anesthesiology Resident, Universidad de Cartagena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Ketofol-001
Record Dates: First submitted 2012-07-02; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Anesthesia; Reaction
Keywords: ketamine; propofol anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketofol 1:1 (Active Comparator): 1. Anesthesia-sedation KETOFOL 1-1: Two milligrams per kilogram of ketamine plus two milligrams per kilogram of propofol in a solution 1:1 (one milligram of ketamine per one milligram of propofol) was given to those patients randomly asigned to this group, who were scheduled for any short surgical procedures previously defined in the inclusion criteria.
  Interventions: Drug: Ketamina-Propofol Combination
- Ketofol 1:2 (Experimental): 2. Anesthesia-sedation KETOFOL 1-2: One milligram per kilogram of ketamine plus two milligrams per kilogram of propofol in a solution 1:2 (one milligram of ketamine per two milligrams of propofol) was given to those patients randomly asigned to this group, who were scheduled for any short surgical procedure previously defined in the inclusion criteria.
  Interventions: Drug: Ketamina-Propofol Combination

INTERVENTIONS:
Drug: Ketamina-Propofol Combination — After randomization to the study group, the patients were given:
  Procedures < 10 minutes
  1. Ketamine-Propofol Combination KETOFOL 1:1
     * Propofol: 0.2 cc/kg (10 mg/cc = 2 mg/kg)
     * Ketamine: cc/kg 0.04 (50 mg/cc = 2 mg/kg)
     * Simple 1% lidocaine: 0,1 cc/kg (10 mg/cc = 1 mg/kg)
  2. Ketamine-Propofol Combination KETOFOL 1:2
     * Propofol: 0.2 cc/kg (10 mg/cc = 2 mg/kg)
     * Ketamine: 0.02 cc/kg (50 mg/cc = 1 mg/kg)
     * Simple 1% lidocaine: 0,1 cc/kg (10 mg/cc = 1 mg/kg)
  Procedures > 10 minutes
  In addition to the initial bolus, an infusion was started:
  KETOFOL 1:1
  20 cc of propofol (10 mg/cc = 200 mg in total) 4 cc of ketamine (50 mg/cc = 200 mg in total) 10cc lidocaine 1% simple (10 mg/cc = 100 mg in total) 66 cc 0.9% SSN
  KETOFOL 1:2
  20 cc of propofol (10 mg/cc = 200 mg in total) 2 cc of ketamine (50 mg/cc = 100 mg in total) 10cc lidocaine 1% simple (10 mg/cc = 100 mg in total) 68 cc 0.9% SSN
  Speed infusion:
  0,03cc/kg/min
  Other Names: Ketofol

SUMMARY:
OBJECTIVE: To determine the efficacy of ketamine-propofol anesthesia in a mixture 1:2 (1 mg of ketamine per 2 mg of propofol) for short minimally invasive surgical procedures.

METHODS: The investigators performed a prospective study through randomization of 77 patients undergoing short surgical procedures in two study groups: one received a mixture of ketamine-propofol in a 1:1 ratio, and the other received a 1:2 mixture. Data were stored in an Excel spreadsheet and analyzed using the statistical program Epi-Info (TM) 3.5.3. The investigators performed the comparison of qualitative and quantitative variables.

KEY WORDS: ketamine, propofol, anesthesia.

DETAILED DESCRIPTION:
In recent years there has been particular interest in ketamine-propofol for sedation of patients who are candidates for short minimally invasive surgical procedures. In some centers in Canada and the U.S. is, in fact, the first choice of sedation in the ED. There are also publications of their usefulness for pediatric procedures, interventional radiology, hematology, oncology, neurosurgery, ophthalmology, orthopedic surgery, CABG, burn patients, gastroenterology, etc.; its benefits as mixed anesthetic technique in patients with neuraxial anesthesia are recognized. Around this, the literature is generous to provide us with evidence to use it in our daily practice.

There is no precise definition of what the ketofolis. Generally refers to the 50:50 mixture of ketamine and propofol, 0.5 mg / kg of each. However, a broader definition considered that ketofol is the combination of ketamine and propofol, regardless of the ratio to each other (the initial dose of each can be scaled up to 3 mg / kg). When they are used in infusion, the dose is 100μg/kg/min.

The combination of ketamine and propofol offers advantages from a theoretical viewpoint, and as already shown, from a clinical standpoint. Ketamine-propofol technique simulates the conditions of general anesthesia because the patient is still unconscious, and although they should be available for when needed, saves anesthetic equipment as endotracheal tubes, laryngeal masks, anesthesia machine, etcetera. Avoid also the risk of malignant hyperthermia by halogenated because the patient is not exposed to pure technical inhalation or balanced techniques. Guitar proposed the ketamine-propofol mixture in 1991, however, was Friedberg who first published his benefits March 26, 1992. Friedberg was based on the technique of Vinnik using ketamine-diazepam for outpatient cosmetic procedures performed in the office. Ketamine is an aryl cyclohexamine (2-0-chlorophenyl-2-methylamino cyclohexanone) synthesized in 1961, with sedative, amnesic and analgesic properties, acting as NMDA receptor antagonist and agonist μ and σ opioid receptors. It starts to act at the first minute after intravenous application. Its duration of action is 15-30 min intravenously; the elimination half-life is 2-3 hours. Is soluble in water and lipophilic, which allows its administration by multiple routes. At low doses is primarily an analgesic and mild sedative, at higher doses produced a catatonic dissociated state which level of sedation is not increased with subsequent doses. Ketamine should be dosed based on ideal body weight and infused in 1 to 2 minutes.

It has been used extensively in health institutions with limitations for patient monitoring or limitations to address advanced airway devices, because it preserves airway reflexes, indeed, patients can swallow even if they are completely dissociated. Ketamine also increases blood pressure and myocardial oxygen demand by stimulating the cardiovascular tone by inhibiting the reuptake of catecholamines centrally. Ketamine is a respiratory stimulant, but may cause transient respiratory depression and even apnea during the first 3 minutes of administration. This problem is most often observed when the drug is administered rapidly or in association with other respiratory depressants such as benzodiazepines. It also produced laryngospasm in 0.4% of a large series of patients, so initially was contraindicated for intraoral procedures, but today it is still used for dental procedures.

Of the 11,589 children in the meta-analysis of Green who were administered ketamine, only 2 (0.017%) required intubation for laryngospasm. Other adverse effects of ketamine include feelings of dissociation from the body, unpleasant dreams, hallucinations or illusions, delusions, etc. Produces electrophysiological dissociation between neocortex, thalamus and limbic system, stimulation of the hippocampus and other subcortical nuclei, or the depression of the visual and auditory nuclei, which would lead to the misperception of external stimuli.

The emergent phenomenon, known as dysphoric reaction on waking from anesthesia induced by ketamine, can occur in up to 20% of cases. Sedatives, counseling and music have proven to reduce the occurrence of these reactions. Vomiting occurs in 5 to 15% of patients emerging from a dissociative state. A rash may appear immediately after injection of ketamine that resolves spontaneously within 20 minutes, and does not use in subsequent administrations. The salivation is a common problem in children so antisialagogues are imperative; this is less common in adults, and the use of antisialagogues may slightly increase the incidence of adverse respiratory events.

In dissociative doses, ketamine produces a reliable analgesia. It is the only intravenous anesthetic with properties such as amnesia, sedation and analgesia that make of ketamine the only intravenous anesthetic that can be used alone to provide anesthesia. However, repetitive use and higher doses induces tolerance. In its favor is the high margin of safety: Strayer & Nelson reviewed over 70000 patients, and only documented one significant cardiorespiratory event attributed to ketamine.

It was felt for a long time that ketamine was contraindicated in patients with traumatic brain injury, but evidence now suggests that those patients may benefit because ketamine preserves cerebral blood flow. Ketamine also elevates intraocular pressure: it should be avoided in patients with glaucoma. Also is contraindicated in psychosis and hyperthyroidism.

The 2.6 diisopropylphenol, also known as propofol, is an alkyl with pure sedative action. It was first used widely as a hypnotic by 1986, achieving great popularity for its rapid onset of action and short half-life effectiveness. Its onset of action is less than one minute and duration of 5 to 15 minutes. It can be administered only by intravenous bolus only for short procedures or infusions for longer procedures. Lean body weight (ideal weight corrected in the morbidly obese) must be used to calculate the initial bolus, and real weight to calculate the maintenance dose.

Propofol is prepared as a lipid emulsion containing soy lecithin and egg, with the potential for allergic reactions in people sensitive to these components. The lipid emulsion promotes bacterial growth, so that the vial must be protected to avoid contamination. The low pH causes burning pain when applied, that is why it is coadministered with lidocaine to reduce pain of injection. Its mechanism of action is based on the potentiation of the GABA receptor activity and sodium channel blockade. Propofol has no analgesic action, so it is necessary to achieve deep sedation for painful procedures, exposing the patient to their respiratory depressant and hypotensive effects (desaturation and apnea) at the doses required to produce adequate sedation. Induces transient hypoxia in the 5 to 20% of patients, and 10-25% decrease in mean arterial pressure. Its use is safe, with a documented need for CPR in 2 of 49,836 patients. Agitation, tachycardia, confusion and hallucinations secondary to the use of propofol can be reversed with the use of physostigmine. There is not agent to reverse the hypnotic effects of propofol.

The combination of ketamine and propofol seeks to limit the adverse effects of each of the two drugs, and synergize their analgesic, hypnotic and sedative effects because they use less dose of each to achieve the same anesthetic and cardiovascular effects. Seven studies support the concept of synergy because similar quality of anesthesia was achieved with lower doses of propofol and ketamine. Propofol is an excellent sedative but has no analgesic effects. Hypotension and respiratory depression of propofol may be offset by the sympathomimetic effects of ketamine. Eight studies confirm the protective effect of ketamine on propofol-induced hypotension. Vomiting and hallucinations of ketamine can be reduced by antiemetic and hypnotic effects of propofol. Propofol reduces dysphoric reactions of ketamine, in some cases to zero.

There have been multiple schemes, dose and proportions in the mixture of ketamine-propofol. Is not entirely clear, however, what proportion of ketamine-propofol is better. Willman and Andolfatto used a proportion 1: 1, meaning that for each mg of ketamine they administered 1 mg of propofol, obtaining satisfactory results for the patient, and highly effective in achieving the therapeutic goal. But our question is if different proportions of this mixture can produce the same sedative benefits with better secondary effects profile. This study was based on a ratio 1:2 (1 mg of ketamine per 2 mg of propofol) compared with a 1:1 ratio mixture in patients who went for short minimally invasive procedures and see if they had fewer adverse effects. Sharieff et al used already ketamine-propofol combination in a 1:2 ratio in a small group of 20 pediatric patients.

MATERIALS AND METHODS

Study Design It was a randomized, controlled, prospective study in patients undergoing minimally invasive procedures of less than an hour. Informed consent was obtained from each of the admitted patients. The study was approved by the ethics committee of the University of Cartagena.

Setting and population The study was conducted in two tertiary care academic institutions. Patients who met selection criteria were randomized (according to a table of random numbers generated on the website: http://stattrek.com/tables/random.aspx) to be assigned to one of the two research groups, between March and September 2011.

Study Protocol During the study period, one researcher was responsible for selecting and inviting patients to be part of the study in the area for the preparation of patients before entering surgery. Once patients nodded in their participation, the informed consent were read and explained, which must be signed before assigning the patient to one of the groups. Later the patient was conducted to the operating room. One anesthesia machine connected to a source of 100% oxygen was available, as well as devices for handling non-invasive and invasive airway (nasal cannula, face masks for all sizes, Guedel cannula, laryngoscope with Macintosh and Miller blades of all sizes, orotracheal tubes of all sizes and laryngeal masks of all sizes). Also there were additional anesthetic drugs in case the anesthesiologist required inducing a deep anesthetic plane, or if required the rapid securing the airway with advanced devices. There was always at least one researcher (senior resident) in the operating room who was on charge of providing the medications, and monitor and record the hemodynamic and respiratory parameters. The researcher was careful to correct any anesthetic complication that arises in the course of surgery.

The following were the inclusion criteria:

1. Patient scheduled for minimally invasive procedures of less than an hour: reduction of dislocations and fractures, lavage and debridement of ulcers, drainage of abscesses, removal of osteosynthesis material, hernia umbilical, thoracotomies, circumcision, curettage, suturing tissue soft, burn care, etc.
2. Patients who have not eaten solid food within 8 hours before, or liquids in the two hours before
3. Be an adult or emancipated minor

The following were the exclusion criteria:

1. An acute lung infection
2. Procedures involving stimulation of the posterior pharynx
3. Coronary heart disease, CHD, and angina or suspected aortic dissection
4. History of uncontrolled hypertension or BP> 140/90mmHg
5. Injury cerebral focal neurological deficit or loss of consciousness
6. Mass in CNS, hydrocephalus or other conditions with increased intracranial pressure.
7. Glaucoma or eye damage
8. History of porphyrias
9. Prior hyperthyroidism or thyroid hormone replacement
10. Pregnancy or lactation Major psychiatric disorder
11. Previous mild allergic reaction to ketamine, propofol, lidocaine, or egg albumin
12. Patient who refuses to provide informed consent

After random assignment to study group, patients were given one of the following two combinations:

1. Anesthesia-sedation KETOFOL 1-1: 1 mg of ketamine per 1 mg of propofol.
2. Anesthesia-sedation KETOFOL 1-2: 1 mg of ketamine per 2 mg of propofol.

Then the duration of the procedure was set to determine whether the patient would require bolus only (patients whose procedure lasted less than 10 minutes) or bolus and infusion (patients whose procedure lasted more than 10 minutes):

<10 minutes

The solution was prepared in a 20 cc syringe with:

KETOFOL 1-1:

* Propofol: 0.2 cc / kg (10mg/cc = 2mg/kg)
* Ketamine: 0.04 cc / kg (50mg/cc = 2mg/kg)
* 1% Lidocaine simple: 0.1 cc / kg (10mg/cc = 1mg/kg)

KETOFOL 1-2:

* Propofol: 0.2 cc / kg (10mg/cc = 2mg/kg)
* Ketamine: 0.02 cc / kg (50mg/cc = 1mg/kg)
* 1% Lidocaine simple: 0.1 cc / kg (10mg/cc = 1mg/kg)

The allocated solution was administered at a minimum of three minutes to reduce to a minimum the incidence of respiratory depression. If the patient did not reach an adequate level of sedation / anesthesia, the patient received additional boluses every three minutes like this:

KETOFOL 1-1:

* Propofol: 0.1 cc / kg (10mg/cc = 1mg/kg)
* Ketamine: 0.02 cc / kg (50mg/cc = 1mg/kg)

KETOFOL 1-2:

* Propofol: 0.1 cc / kg (10mg/cc = 1mg/kg)
* Ketamine: 0.01 cc / kg (50mg/cc = 0.5 mg / kg)

> 10 minutes

These patients also required the initial bolus, and then an infusion of the same mixture of drugs started. The bolus dose was prepared similarly to as described above, and infusion solutions were prepared as follows:

KETOFOL 1-1:

In a volume of 100cc:

* 20 cc of propofol (10mg/cc = 200mg total)
* 4 cc of ketamine (50mg/cc = 200mg total)
* 10 cc 1% lidocaine simple (10mg/cc = 100 mg total)
* 66 cc 0.9% SSN

KETOFOL 2-1:

In a volume of 100cc:

* 20 cc of propofol (10mg/cc = 200mg total)
* 2 cc of ketamine (50mg/cc = 100mg total)
* 10 cc 1% lidocaine simple (10mg/cc = 100 mg total)
* 0.9% SSN 68 cc

The volumes administered were as follows:

Ketofol 1-1:

Bolus in three minutes and immediately begins the infusion to 0.03 cc / kg / min (60 μgr / kg / min of ketamine + 60 μgr / kg / min of propofol).

Ketofol 1-2:

Bolus in three minutes and immediately begins the infusion to 0.03 cc / kg / min (30 μgr / kg / min of ketamine + 60 μgr / kg / min of propofol).

The infusions were suspended 5 minutes before the end of the surgical procedure.

The data were stored in a Microsoft Excel spreadsheet for tabulation and analysis by one of the researchers behind the study.

Measurements The doses of the drugs used were administered by ideal weight corrected (ideal weight + 40% of the difference between actual weight and ideal weight). The satisfaction of patients and surgeons was evaluated in a 5-item scale: extremely satisfied, very satisfied, neither satisfied nor dissatisfied, dissatisfied and very dissatisfied. Sedation / analgesia was considered successful if the procedure was completed without the need for other anesthetic drugs different from the protocol, and no adverse effects obliged the suspension of the procedure. Apnea was defined as cessation of breathing for at least 20 seconds. Hypotension was defined as 20% decrease in mean arterial pressure. Bradycardia was defined as a pulse of less than two standard deviations below normal values defined by the American Heart Association (AHA_ for its acronym in Ingles_). Hypoxia was defined by an oxygen saturation of less than 90%.

Data Analysis Data were analyzed using Epi-Info (TM) 3.5.3.

LIMITATIONS

Within the constraints of the study is the limited sample size could have influenced the study's inability to achieve statistical significance in the differences obtained for most of the evaluated parameters between the two groups. Ketofol was not compared with other regimens of sedation, analgesia, and therefore cannot make any representations regarding its safety and efficacy faced with other schemes. The study was not applied to the pediatric population, which responds favorably to the administration of ketamine. Adverse effect was recorded as any manifestation of agitation, pain, nausea, etc., regardless of severity, which may exaggerate the incidence of adverse events of ketamine-propofol combination.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for minimally invasive procedures less than an hour to complete: reduction of dislocations and fractures, lavage and debridement of ulcers, drainage of abscesses, removal of osteosynthesis material, hernia umbilical, thoracotomies, circumcision, curettage, suturing tissue soft, burn care, etc.
2. Patients who have not eaten solid food within 8 hours before or liquids in the two hours before
3. Be an adult or emancipated minor

Exclusion Criteria:

1. An acute lung infection
2. Procedures involving stimulation of the posterior pharynx
3. Coronary heart disease, CHD, and angina or suspected aortic dissection
4. History of uncontrolled hypertension or BP > 140/90mmHg
5. Injury cerebral focal neurological deficit or loss of consciousness
6. Mass in CNS, hydrocephalus or other conditions with increased intracranial pressure.
7. Glaucoma or eye damage
8. History of porphyrias
9. Prior hyperthyroidism or thyroid hormone replacement
10. Pregnancy or lactation Major psychiatric disorder
11. Previous mild allergic reaction to ketamine, propofol, lidocaine, or egg albumin
12. Patient who refuses to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
EFFICACY OF KETAMINE-PROPOFOL FOR SHORT SURGICAL PROCEDURES | 7 months
  Sedation / analgesia was considered successful if the procedure was completed without the need for other anesthetic drugs are different from the protocol, and yes no adverse effects to oblige the completion of the procedure. Apnea was defined as cessation of breathing for at least 20 seconds. Hypotension was defined as 20% decrease in mean arterial pressure. Bradycardia was defined as a pulse of less than two standard deviations below normal values defined by the American Heart Association (AHA_ for its acronym in Ingles_). Hypoxia was defined by an oxygen saturation of less than 90%.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Poveda, Resident, Principal Investigator — University of Cartagena